CLINICAL TRIAL: NCT05260580
Title: Application of Empowerment Strategies for Gender Equality Among Nursing Students in In-service Education
Brief Title: Application of Empowerment Strategies for Gender Equality Among Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Chia Jung Hsieh, Ph.D., RN, Associate Professor, National Taipei University of Nursing and Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FJU-IRB C109027
Record Dates: First submitted 2022-02-18; First posted 2022-03-02 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Gender Equality
Keywords: Medical system; gender equality; gender training; gender sensitivity

STUDY DESIGN:
Intervention Model Description: one group (Experiment group)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Two-hour sessions per week for 18 weeks (Experimental): The classroom learning of study subjects and clinical care experience of in-service students are both very important in this intervention course. The teaching method will primarily focus on empowerment strategies, with support from the school's digital action learning platform for teaching-related activities.
  Interventions: Other: No Intervention: Routine care

INTERVENTIONS:
Other: No Intervention: Routine care

SUMMARY:
Gender mainstreaming is a global development trend, as gender disparity has an impact on the development of the social, economic, political, and medical ecologies, as well as people's lives. Understand that gender education involves systematic and structured planning to break students' gender blindness. And to implement health and gender as essential foundations of human rights. Educators need to use systematic curriculum planning and design to conduct gender impact assessments on current curriculum, plans, or policies in the field of health care, so as to strengthen learners' analysis of health problems and consider gender factors at the same time. It is necessary to guide students to incorporate gender perspectives into their thinking so as to help students adopt diversified problem-solving strategies and actions in the care process.

This study used a quasi-experimental research design. The students of a university nursing department were the research subjects. We had a total of 44 participants through a convenient sampling method (one class per week, two hours each time, for a total of 18 weeks). At the same time, we collected the subject's learning reflections on gender issues and conducted the content analysis. The gender stereotype and role attitude scale were used as instruments, and the data were analyzed by the paired t-test method using the software package SPSS 21.0. The research results showed that through the concept of empowerment, students can be enlightened about their gender concepts, explicit knowledge can be transformed into tacit knowledge, and the empowerment process can prompt individuals to truly understand, apply knowledge, and start from the subject experience of learning, also transforming their learning experience. Individuals can become aware of their behaviors, thereby generating problem-solving abilities and practical actions with the gender perspective.

DETAILED DESCRIPTION:
Gender mainstreaming is an important international trend, and staff in the health care system are also affected by this trend, and jointly advocate for the implementation of gender sensitivity in the medical care field. Therefore, it is understood that the promotion of gender education requires systematic and structural planning to break the gender blindness of students and to implement health and gender as an important basis for human rights.

Educators need to use systematic curriculum planning and design to conduct gender impact assessments on current curriculum, plans, or policies in the field of health care, so as to strengthen learners' analysis of health problems and consider gender factors at the same time. It is necessary to guide students to incorporate gender perspectives into their thinking so as to help students adopt diversified problem-solving strategies and actions in the care process.

This study used a quasi-experimental research design. The students of a university nursing department were the research subjects. We had a total of 44 participants through a convenient sampling method (one class per week, two hours each time, for a total of 18 weeks). At the same time, we collected the subject's learning reflections on gender issues and conducted the content analysis. The gender stereotype and role attitude scale were used as instruments, and the data were analyzed by the paired t-test method using the software package SPSS 21.0. The research results showed that through the concept of empowerment, students can be enlightened about their gender concepts, explicit knowledge can be transformed into tacit knowledge, and the empowerment process can prompt individuals to truly understand, apply knowledge, and start from the subject experience of learning, also transforming their learning experience. Individuals can become aware of their behaviors, thereby generating problem-solving abilities and practical actions with the gender perspective.

ELIGIBILITY:
Inclusion Criteria:

* Students in a university nursing department (third year students) who have taken two credits of "Gender and Health Care" as an elective in a specific in-service class will be the study object of this project, as determined by a suitable sampling procedure.

Exclusion Criteria:

* Students that have selected "Gender and Health Care" but do not wish to participate in this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
The scale of Gender Role Stereotype | Baseline, pre-intervention(T0)
  The scale of Gender Role Stereotype Gender role stereotypes in the areas of personality traits, occupation, family issues, activities, and games are grouped into the theme dimensions of the questionnaire. For each item, there are three options. If the options are appropriate for both boys and girls, 1 point will be awarded; otherwise, no points will be awarded.
The scale of Gender Role Attitudes Scale | Baseline, pre-intervention(T0)
  The scale of Gender Role Attitudes Scale Gender role attitude questions, a total of six questions, according to the four levels of strongly disapprove, disapprove, agree, and strongly agree, designated as 1, 2, 3, and 4 points respectively, the higher the score, the more inclined to gender equality, autonomy, non-traditional gender role attitudes.
The scale of Gender Role Stereotype | eighteen weeks after intervention(T1)
  The scale of Gender Role Stereotype Gender role stereotypes in the areas of personality traits, occupation, family issues, activities, and games are grouped into the theme dimensions of the questionnaire. For each item, there are three options. If the options are appropriate for both boys and girls, 1 point will be awarded; otherwise, no points will be awarded.
The scale of Gender Role Attitudes Scale | eighteen weeks after intervention(T1)
  The scale of Gender Role Attitudes Scale Gender role attitude questions, a total of six questions, according to the four levels of strongly disapprove, disapprove, agree, and strongly agree, designated as 1, 2, 3, and 4 points respectively, the higher the score, the more inclined to gender equality, autonomy, non-traditional gender role attitudes.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Jung Hsieh, PhD, Study Director — 365,Ming-te Road,Peitou District,Taipei City
Locations (1):
- National Taipei University of Nursing and Health Sciences, Taipei, Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bandura A. Self-efficacy: toward a unifying theory of behavioral change. Psychol Rev. 1977 Mar;84(2):191-215. doi: 10.1037//0033-295x.84.2.191. No abstract available. PMID 847061
- [Result] Cheng LF, Yang HC. Learning about gender on campus: an analysis of the hidden curriculum for medical students. Med Educ. 2015 Mar;49(3):321-31. doi: 10.1111/medu.12628. PMID 25693991
- [Result] Anthony AS. Gender bias and discrimination in nursing education: can we change it? Nurse Educ. 2004 May-Jun;29(3):121-5. doi: 10.1097/00006223-200405000-00011. PMID 15167580
- [Result] Dyck JM, Oliffe J, Phinney A, Garrett B. Nursing instructors' and male nursing students' perceptions of undergraduate, classroom nursing education. Nurse Educ Today. 2009 Aug;29(6):649-53. doi: 10.1016/j.nedt.2009.02.003. Epub 2009 Mar 6. PMID 19269071
- [Result] Forneris SG, Peden-McAlpine C. Evaluation of a reflective learning intervention to improve critical thinking in novice nurses. J Adv Nurs. 2007 Feb;57(4):410-21. doi: 10.1111/j.1365-2648.2007.04120.x. PMID 17291205
- [Result] Hawks JH. Organizational culture and faculty use of empowering teaching behaviors in selected schools of nursing. Nurs Outlook. 1999 Mar-Apr;47(2):67-73. doi: 10.1016/s0029-6554(99)90071-4. No abstract available. PMID 10227032
- [Result] Kuokkanen L, Leino-Kilpi H, Numminen O, Isoaho H, Flinkman M, Meretoja R. Newly graduated nurses' empowerment regarding professional competence and other work-related factors. BMC Nurs. 2016 Mar 24;15:22. doi: 10.1186/s12912-016-0143-9. eCollection 2016. PMID 27013927
- [Result] Macintosh J. Gender-related influences in nursing education. J Prof Nurs. 2002 May-Jun;18(3):170-5. doi: 10.1053/jpnu.2002.125475. PMID 12096366
- [Result] Meadus RJ, Twomey JC. Men student nurses: the nursing education experience. Nurs Forum. 2011 Oct-Dec;46(4):269-79. doi: 10.1111/j.1744-6198.2011.00239.x. PMID 22029770
- [Result] Moore SC, Ward KS. Nursing Student Perceptions of Structural Empowerment. Nurs Educ Perspect. 2017 Jan/Feb;38(1):32-33. doi: 10.1097/01.NEP.0000000000000096. PMID 29194241
- [Result] Park S, Kwon DW, Kim D, Kim SH. Influences of gender-related perceptions and experiences on nursing professionalism: A cross-sectional study. Nurs Health Sci. 2019 Dec;21(4):515-522. doi: 10.1111/nhs.12636. Epub 2019 Aug 30. PMID 31469236
- [Result] Reitinger E, Lehner E, Pichler B, Heimerl K. ["Doing gender" in a nursing home for the elderly : Perspectives of staff and management]. Z Gerontol Geriatr. 2016 Dec;49(8):700-705. doi: 10.1007/s00391-016-1147-5. Epub 2016 Oct 28. German. PMID 27796518